CLINICAL TRIAL: NCT02853318
Title: A Phase II Evaluation of Pembrolizumab in Combination With IV Bevacizumab and Oral Metronomic Cyclophosphamide in the Treatment of Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Pembrolizumab, Bevacizumab, and Cyclophosphamide in Treating Patients With Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 270715; NCI-2016-00534 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 270715 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Serous Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Undifferentiated Fallopian Tube Carcinoma; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab, bevacizumab, cyclophosphamide) (Experimental): Patients receive pembrolizumab IV over 30 minutes and bevacizumab IV over 30-90 minutes on day 1 and cyclophosphamide PO QD on days 1-21. Treatment repeats every 3 weeks for up to 17 courses in the absence of disease progression or unacceptable toxicity. Patients without evidence of disease progression may continue treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies the combination of pembrolizumab, bevacizumab, and low dose oral cyclophosphamide in treating patients with recurrent ovarian, fallopian tube, or primary peritoneal cancer. Monoclonal antibodies, such as pembrolizumab and bevacizumab, may block tumor growth in different ways such as boosting your own immune system to find, recognize and kill tumor cells as well as by blocking the growth of new blood vessels necessary for tumor growth and nutrition. Drugs used in chemotherapy, such as low dose oral cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, as well as by further enhancing your own body's immune response against cancer cells. As these three drugs have all been shown to improve the immune response against cancer cells giving pembrolizumab, bevacizumab, and cyclophosphamide together may work better in treating patients with recurrent ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate improvement in progression-free survival for patients treated with anti-programmed cell death 1 (anti-PD1) pembrolizumab in combination with intravenous (IV) bevacizumab and oral metronomic cyclophosphamide as compared to patients treated with other second line chemotherapeutic agents.

SECONDARY OBJECTIVES:

I. To obtain pilot data on clinical response rates using both Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and immune related response criteria (irRECIST).

II. To obtain data on changes in tumor microenvironment prior to and subsequent to therapy and, to screen for potential biomarkers to predict clinical benefit.

III. To determine the safety and tolerability of the treatment combination in the study population.

IV. To evaluate overall survival in patients treated with anti-PD1 pembrolizumab in combination with IV bevacizumab and oral metronomic cyclophosphamide.

V. To assess the impact of the combination of anti-PD1 pembrolizumab, IV bevacizumab and oral metronomic cyclophosphamide on anti-tumor immune responses in ovarian cancer.

OUTLINE:

Patients receive pembrolizumab IV over 30 minutes and bevacizumab IV over 30-90 minutes on day 1 and cyclophosphamide orally (PO) once daily (QD) on days 1-21. Treatment repeats every 3 weeks for up to 12 months (or 17 courses) in the absence of disease progression or unacceptable toxicity. Patients without evidence of disease progression may continue treatment in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for 1 year, and every 12 weeks and 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have measurable disease per RECIST 1.1 criteria present
* Participant may have serous, endometrioid, clear cell, mucinous or undifferentiated type of recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer

  * Histologic confirmation of the original primary tumor is required via the pathology report
* Participant can be either platinum-sensitive (platinum free interval [PFI] >= 6 months prior to recent recurrence) or platinum-resistant (PFI < 6 months prior to recent recurrence). If the participant has a platinum sensitive disease, she may only enroll in this clinical trial if there is a contraindication for her to receive further treatment with platinum-based chemotherapy (such as serious, persistent toxicity or sever hypersensitivity to platinum agents or she declines standard of care).
* Participant must be willing to undergo core or excisional biopsy of a tumor lesion within 4 weeks (28 days) prior to initiation of treatment on day 1 and after 3 cyles of study treatment; participants for whom newly obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the principal investigator
* Absolute neutrophil count (ANC): >= 1,500 /mcL
* Platelets: >= 100,000 / mcL
* Hemoglobin: >= 9 g/dL or 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine: =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 mL/min for participant with creatinine levels > 1.5 X institutional ULN; glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)
* Urine protein creatine ratio (UPCR) < 1 prior to enrollment
* Serum total bilirubin: =< 1.5 X ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase[SGOT]) and alanine transaminase (ALT) (serum glutamic pyruvic transaminase [SGPT]): =< 2.5 X ULN OR =< 5 X ULN for participants with liver metastases
* Albumin: > 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT): =< 1.5 unless participant is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT): =< 1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Participants of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year); should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Participant has recovered from toxicities of prior chemotherapy or other therapy (to grade 2 or less)
* Participant may have received prior investigational therapy (including immune therapy)
* Participant may have received prior hormonal therapy
* Participant may have received bevacizumab (or other antiangiogenic agent) and/or cyclophosphamide in the past
* Participant has had at least 4 weeks of postoperative recovery from surgery prior to enrollment to ensure complete wound healing; participants with bowel resections at surgery should begin protocol at least 42 days after surgery
* Ability to swallow and retain oral medication
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment or, is taking any other medication that might affect immune function
* Has a known history of active bacillus tuberculosis (TB)
* Hypersensitivity to bevacizumab, cyclophosphamide, pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: participants with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy and, has to be at least 28 days after the surgery
* Has a known additional malignancy that is progressing or requires active treatment: exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or cervical cancer in situ that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 6 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-programmed cell death 1 ligand 1 (PD-L1), or anti-programmed cell death 1 ligand 2 (PD-L2) agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines, and are not allowed
* Active or history of inflammatory bowel disease (colitis, Crohn's), diverticulitis, irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea; active or history of systemic lupus erythematosus or Wegener's granulomatosis
* Participant has clinical symptoms or signs of partial or complete gastrointestinal obstruction or, requires parenteral hydration and/or nutrition
* Participant requires, or is likely to require, more than a two-week course of corticosteroids for intercurrent illness; participant must complete the course of corticosteroids 2 weeks before screening to meet eligibility
* Participant has a serious, non-healing wound, ulcer, or bone fracture
* Participant has a clinically significant cardiovascular disease including:

  * Uncontrolled hypertension, defined as systolic > 150 mmHg or diastolic > 90 mmHg
  * Myocardial infarction or unstable angina within 6 months prior to enrollment
  * New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Participant has a grade II or greater peripheral vascular disease
  * Participant has a clinically significant peripheral artery disease (e.g. those with claudication, within 6 months)
* Participant has organ allografts
* Participant is receiving medication(s) that might affect immune function
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Rosario SR, Long MD, Chilakapati S, Gomez EC, Battaglia S, Singh PK, Wang J, Wang K, Attwood K, Hess SM, McGray AJR, Odunsi K, Segal BH, Paragh G, Liu S, Wargo JA, Zsiros E. Integrative multi-omics analysis uncovers tumor-immune-gut axis influencing immunotherapy outcomes in ovarian cancer. Nat Commun. 2024 Dec 5;15(1):10609. doi: 10.1038/s41467-024-54565-8. PMID 39638782
- [Derived] Zsiros E, Lynam S, Attwood KM, Wang C, Chilakapati S, Gomez EC, Liu S, Akers S, Lele S, Frederick PJ, Odunsi K. Efficacy and Safety of Pembrolizumab in Combination With Bevacizumab and Oral Metronomic Cyclophosphamide in the Treatment of Recurrent Ovarian Cancer: A Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2021 Jan 1;7(1):78-85. doi: 10.1001/jamaoncol.2020.5945. PMID 33211063

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide)
Started | 40
Completed | 39
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38
  Black | 0
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 40
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead
  Participants
    0 | 28
    1 | 12
BRCA mutation status [Count of Participants; unit: Participants] — The mutation status includes germline and somatic mutations.
  Participants
    positive | 14
    negative | 23
    unknown | 3
Baseline PDL1 expression [Count of Participants; unit: Participants]
  positive | 19
  negative | 17
  unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events Assessed by Common Terminology Criteria for Adverse Events
Description: The highest observed adverse event will be tabulated by grade across all dose levels and cycles.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 40
Participants
  No Adverse Events | 1
  Grade I | 9
  Grade II | 20
  Grade III | 9
  Grade IV | 1
  Grade V | 0

2. Primary Outcome: Progression-free Survival (PFS)
Description: Will be summarized using standard Kaplan-Meier methods, with estimates of median survival and given survival rates will be obtained with 90% confidence intervals.
Time Frame: Time from the start of the study treatment until PFS event, assessed up to 1 year after the last subject enrolls
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 40
months | 10.0 [6.5 to 17.4]

3. Secondary Outcome: Duration of Overall Survival
Description: as for outcome 2
Time Frame: Up to 1 year after enrollment of the last subject
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 40
months | 16.0 [12.5 to 26.1]

4. Secondary Outcome: An Anti-tumor Immune Response in Circulation and Tumor Tissue
Description: Assessed with immunohistochemistry (IHC), Nannostring, Flow Cytometry and Luminex assay.
Time Frame: Up to 1 year
Population: The IHC, Nannostring, Flow Cytometry and Luminex assays were not completed.
Arm/Group | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 0

5. Secondary Outcome: Objective Tumor Response Assessed by Modified RECIST Version 1.1 Criteria
Description: Frequency of response will be summarized with a 90% confidence interval.
  An objective response is defined as a CR or PR, while a non-responder is defined as a SD or PD.
Time Frame: Up to 6 months after enrollment start of treatment
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide)
Number analyzed (Participants) | 40
proportion of participants | 0.475 [0.349 to 0.603]

ADVERSE EVENTS:
Time Frame: Adverse Events: Through study completion up to 3 years.
Arm/Group | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide)
All-Cause Mortality (participants affected / at risk) | 27/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 38/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Bevacizumab, Cyclophosphamide) (N=40)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (4)
Eye pruritus (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 14 (20)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (10)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 16 (20)
Feeling cold (General disorders) | 2 (2)
Influenza like illness (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 5 (7)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood creatine increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (11)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (4)
Urine analysis abnormal (Investigations) | 1 (1)
Urine protein/creatinine ratio increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 5 (8)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Taste disorder (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Hypertension (Vascular disorders) | 14 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT02853318/Prot_SAP_000.pdf